CLINICAL TRIAL: NCT03783806
Title: Postural Control in Degenerative and Inflammatory Diseases of the Hip
Acronym: PCHOAI
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Szeged University (Other)
Responsible Party: Principal Investigator, Edit Nagy, PhD, Head of Unit, Szeged University
Other Study IDs: PCHOAI
Record Dates: First submitted 2018-12-19; First posted 2018-12-21 (Actual); Last update posted 2018-12-24 (Actual); Status verified 2018-12

CONDITIONS: Hip Osteoarthritis; Hip Arthritis
Keywords: hip, postural control, degenerative, inflammation
MeSH Terms: conditions — Osteoarthritis, Hip; Inflammation

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Osteoarthrosis (OA): Patients with primary osteoarthrosis, waiting for a total hip replacement. Determination of functional status, posturography measurements, postural tests.
  Interventions: Diagnostic Test: Posturography measurements
- Rheumatoid arthritis (RA): Patients with rheumatoid arthritis affecting hip joint. Determination of functional status, posturography measurements, postural tests.
  Interventions: Diagnostic Test: Posturography measurements
- Control (C): The healthy reference group was matched with the patient groups for age, gender and body mass index (BMI). Determination of functional status, posturography measurements, postural tests.
  Interventions: Diagnostic Test: Posturography measurements

INTERVENTIONS:
Diagnostic Test: Posturography measurements — Determination of functional status, Posturography measurements, postural tests

SUMMARY:
Patients with primary hip osteoarthritis (OA group) and patients with inflammatory hip disease (RA group) and healthy subjects (control group) are enrolled in the study. The aim of our study is to determine the postural control in patients suffering from OA and RA of the hip joint during different conditions, i.e., on both stable and compliant surfaces with opened or closed eyes to determine the possible differences between these two diseases in this respect.

DETAILED DESCRIPTION:
Determination of functional status, using the following outcome measures: Harris Hip Score, the Functional status of the hip joint is rated with the Harris Hip Score (HHS), Visual Analogue Scale, Western Ontario and McMaster Universities Osteoarthritis Index, Timed Up & Go test.

Posturography measurements, Postural control tests

The Clinical Test of Sensory Interaction on Balance (CTSIB) uses different conditions to test how people adapt to changing sensory conditions during the maintenance of stance. We used the modified CTSIB by NeuroCom to perform the test on a computerized force plate to measure the body sway. Static postural stability [displacement of Centre of Pressure (CoP)] was measured during standing on a single force platform (Stabilometer, ZWE-PII) for 20-s periods in a quiet room. Signals were amplified and sampled at 16 Hz via an analogue-to-digital converter. Subjects stood barefoot on the platform, with the feet positioned side by side and arms hanging freely at their side. Toe-out was positioned to subjects' comfort. The CoP excursions along antero-posterior (AP) and medio-lateral (ML) axes were performed both on firm (the stable surface of the platform) and foam surfaces [an Airex Balance Pad (dimensions: 50 cm length x 41 cm width x 6 cm height) placed on the platform], always starting with standing on the stable surface. In each condition, subjects had to stand first with the eyes open (EO), when subjects had to look at a target fixed at eye level at a distance of approximately 1 m, and then measurements were also performed with closed eyes (EC).

ELIGIBILITY:
Inclusion Criteria:

* C-reactive protein and Westergreen values had to be under the upper level of the normal values.
* Patients should have unilateral hip pain on most of the days for several months
* Controls should have no hip pain or functional impairment in the hip joint or any other joint of the lower extremities.

Exclusion Criteria:

* history of trauma to the hip joint or in the pelvic region,
* previous hip fracture or hip surgery,
* hip joint infection and congenital or developmental diseases
* any complaints in the other joints of the lower limbs
* any disease that could worsen their physical or balance parameters
* cancer,
* endocrine,
* cerebrovascular disease,
* Parkinson's syndrome,
* epilepsy,
* polyneuropathy,
* neuromuscular disorder,
* cardiovascular disease without medication,
* atherosclerosis of the lower extremities

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Patients with primary hip osteoarthritis (OA group), patients with inflammatory hip disease (RA group) and healthy subjects (control group) are enrolled in the study. All subjects were independent and capable of self-care and daily household tasks.
Sampling Method: Probability Sample
Enrollment: 90 (Estimated)
Dates: Start 2015-01-01 (Actual); Primary Completion 2018-12-18 (Actual); Study Completion 2018-12-18 (Estimated)

PRIMARY OUTCOMES:
Harris Hip Score (HHS) | 1 hour
  The score has a maximum at 100 points (best possible function), covering pain (part I, 1 item, 0-44 points), function and activities (part II, 7 items, 0-47 points) and range of motion and absence of deformity (part III, 3 items, 0-9 points). [Grading: <70 poor, 70-79 fair, 80-89 good, 90-100 excellent
Visual Analogue Scale | 1 hour
  Hip pain (average pain on movement over the previous 72 hours) is assessed by using a Visual Analogue Scale (VAS) (the range of the scale: 0-100 mm; where the subjects subjectively judge the actual level of pain between the minimum and maximum range. The meaning of the end-points: minimum: no pain- maximum: unbearable pain). The lower values represent better outcome.
Western Ontario and McMaster Universities Osteoarthritis Index | 1 hour
  The Western Ontario and McMaster Universities Osteoarthritis Index (WOMAC) is used to assess pain (WOMAC A, 5 items), joint stiffness (WOMAC B, 2 items) and disability (WOMAC C, 17 items) by using visual analogue scales. Lower scores indicated less pain, less stiffness or less disability.
Timed Up & Go test | 1 hour
  To assess the functional mobility of the subjects, we applied the Timed Up & Go (TUG) test. During the testing procedure, subjects were timed (recorded in seconds) for standing up from a chair (45 cm), walking 3 m, passing around an object and then returning to sitting position in the chair. The subjects were instructed to walk as quickly as possible but not to run. The subjects had three trials with 1 min pause between each trial; the trials were recorded in seconds.
Posturography measurements | 1 hour
  The Clinical Test of Sensory Interaction on Balance (CTSIB) uses different conditions to test how people adapt to changing sensory conditions during the maintenance of stance. We used the modified CTSIB by NeuroCom to perform the test on a computerized force plate to measure the body sway. Static postural stability [displacement of Centre of Pressure (CoP)] was measured during standing on a single force platform (Stabilometer, ZWE-PII) for 20-s periods in a quiet room.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Szeged, Faculty of Health and Social Studies, Department of Physiotherapy, Szeged, Csongrád megye, Hungary

IPD SHARING:
Plan to Share IPD: Undecided